CLINICAL TRIAL: NCT00767871
Title: Changes of Cerebral Glucose Metabolism Associated With the Fear Network Activity Before and After 12 Weeks of Escitalpram Treatment in Panic Disorder
Brief Title: Changes of Cerebral Glucose Metabolism and After 12 Weeks of Escitalpram Treatment in Panic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Bum-Hee Yu, M.D. Ph.D. / Professor, Department of Psychiatry, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SMCIRB2007-01-024; NCT00461383 (obsolete NCT alias)
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Panic Disorder
Keywords: Panic disorder; PET; Escitaopram
MeSH Terms: conditions — Panic Disorder | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escitalopram (Experimental): escitalopram (10-20mg) to panic patients
  Interventions: Drug: Lexapro

INTERVENTIONS:
Drug: Lexapro — 12 week treatment with lexapro

SUMMARY:
Panic disorder is one of the most prevalent psychiatric disorders and recently abnormal fear network is known to be implicated in the pathophysiology of panic disorder. The fear network involves many brain regions such as amygdala, hippocampus, periaqueductal gray (PAG), locus coeruleus, parahippocampal gyrus, frontal cortex, and thalamus. Escitalopram, a highly selective serotonin reuptake inhibitor, is usually effective for panic dis order, but there is little information on how escitalopram affects the fear network.

The specific aim of this study is to test the following hypotheses using 18F-FDG positron emission tomography (PET)

1. Patients with panic disorder will show abnormal activity of the fear network compared to healthy comparison subjects.
2. Patients with panic disorder will show normalized activity of the fear network after 12-weeks of treatment with escitalopram.
3. The changes of fear work after the treatment will be associated with psychological variables and neurohormones.

ELIGIBILITY:
Inclusion Criteria:

* panic disorder
* 20-60 years

Exclusion Criteria:

* history of major psychosis (schizophrenia or bipolar disorder), social phobia, obsessive-compulsive disorder, and generalized anxiety disorder, and posttraumatic stress disorder. The acceptable score on the 17-item Hamilton Depression Rating Scale at entry into the study will be less than 17.
* patients and volunteers with alcohol dependence and current regular use of benzodiazepines will be excluded. Subjects with current or previous regular use of benzodiazepines will be excluded.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2007-03; Primary Completion 2007-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
18FDG-PET, PDSS & HAM-A | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bum-Hee Yu, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea